CLINICAL TRIAL: NCT03061851
Title: A Multicenter, Prospective, Randomized, Controlled Clinical Trial of the Individualized Behavioral Intervention of Smartphone App in the Treatment of Type 2 Diabetes Mellitus
Brief Title: The Individualized Behavioral Intervention of Smartphone App in the Treatment of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Zhixin Health Technology Co., Ltd. (Other)
Collaborators: H & J CRO International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APP20160212
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The enrolled patients will be randomly divided into two groups: the trial group and the control group. The estimated sample size was 200 patients for each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Experimental): given conventional hypoglycemic drug treatment, the treatment plan by the investigators according to the patient's condition may be, this study does not interfere.
  Interventions: Behavioral: conventional treatment
- conventional treatment + maltose app (Experimental): the patients were treated with conventional hypoglycemic drugs. The treatment plan was decided by the investigators according to the patient's condition. The intervention was not done in this study.And joint: maltose App intervention.
  Interventions: Behavioral: conventional treatment; Other: Maltose app

INTERVENTIONS:
Behavioral: conventional treatment — the treatment plan by the investigators according to the patient's condition may be, this study does not interfere.
Other: Maltose app — 1. Weekly diabetes-related science articles.
  2. Patients reported hypoglycemia or other adverse reactions, the competent physician to deal with.
  3. Questionnaires published out the hospital (2 weeks 1), the feedback for the problem.
  4. monitoring of abnormal blood glucose data or the presence of related discomfort, can communicate with the competent physician online.
  5. Personalize the development of diet, exercise program.
  6. different insulin and oral hypoglycemic drug medication time to remind.
  7. hypoglycemic drug side effects query.
  Arms: conventional treatment + maltose app

SUMMARY:
The patients with type 2 diabetes who underwent routine hypoglycemic agents and insulin therapy were evaluated for 48 weeks with maltose software.

DETAILED DESCRIPTION:
This study enrolled 400 patients with type 2 diabetes in five centers in Shandong Province, China. Patients with type 2 diabetes who met the inclusion / exclusion criteria were randomly assigned to the trial group (conventional treatment + maltose app) or the control group (conventional treatment) in a 1: 1 ratio.

The control group: given conventional hypoglycemic drug treatment, the treatment plan by the investigators according to the patient's condition may be, this study does not interfere.

The trial group: the patients were treated with conventional hypoglycemic drugs. The treatment plan was decided by the researcher according to the patient's condition. The intervention was not done in this study.

Interventions include:

1. Weekly diabetes-related science articles.
2. Patients reported hypoglycemia or other adverse reactions, the competent physician to deal with.
3. Questionnaires published out the hospital (2 weeks 1), the feedback for the problem.
4. monitoring of abnormal blood glucose data or the presence of related discomfort, can communicate with the competent physician online.
5. Personalize the development of diet, exercise program.
6. different insulin and oral hypoglycemic drug medication time to remind.
7. hypoglycemic drug side effects query.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients diagnosed with type 2 diabetes, age ≥ 18 years and ≤ 65 years;
2. diagnosis of type 2 diabetes ≥6 months;
3. The patient signed an informed consent form and agreed to collect the data. The trial group agreed to apply the maltose app during the trial period to study popular science articles, to receive software reminders and to answer questions regularly;
4. HbA1c≥7.0% in the last one (≤3 months) before enrollment;
5. be able to use Mobile App;
6. The mobile phone used by the patient must support maltose App installation.
7. Receiving regular diabetes education in the hospital.

Exclusion Criteria:

1. Has participated in any randomized controlled clinical study;
2. To long-term use of insulin pump as the main treatment of type 2 diabetes;
3. patients with type 1 diabetes;
4. pregnant or lactating women;
5. doctor, alcohol, drug abuse, schizophrenia, severe vision and hearing impaired;
6. Can not accept software manager;
7. Other investigators considered it inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with HbA1c <7% after 48 weeks of maltose software intervention | 48 weeks

SECONDARY OUTCOMES:
The changes of HbA1c at baseline, 48 weeks, 36 weeks, 24 weeks and 12 weeks after intervention were compared. | 48 weeks, 36 weeks, 24 weeks and 12 weeks.
The changes of FPG and 2hPG, blood lipids and uric acid in the 48 weeks and 24 weeks after the intervention were compared. | 48 weeks and 24 weeks
The proportion of the different subgroups patients(baseline BMI<24kg/m2, ≥24kg/m2 and ≤28kg/m2 and >28kg/m2; baseline HbA1c≤8%,>8% and ≤10% and >10%) with HbA1c<7% after 48 weeks and 24 weeks of intervention | 48 weeks and 24 weeks
The changes of body weight, waist circumference and hip circumference were compared with baseline at 48 weeks, 36 weeks, 24 weeks and 12 weeks after the intervention. | 48 weeks, 36 weeks, 24 weeks and 12 weeks
The total score of the Morisky compliance questionnaire at baseline, 48 weeks, 36 weeks, 24 weeks, and 12 weeks after intervention was compared with baseline. | 48 weeks, 36 weeks, 24 weeks, and 12 weeks
The total score of self - rating anxiety scale at 48 weeks after intervention was higher than baseline. | 48 weeks
The scores of self - management behavior of patients with diabetes at baseline, 48 weeks, 36 weeks, 24 weeks and 12 weeks after intervention were compared. | 48 weeks, 36 weeks, 24 weeks and 12 weeks
The total score of Kessler's psychological distress scale after 48 weeks of intervention was higher than baseline. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, Study Director — Qingdao Zhixin Health Technology Co., Ltd.
Locations (1):
- Qingdao University Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No